CLINICAL TRIAL: NCT06580041
Title: Precision Care for Major Depressive Disorder
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-41815
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder; Depression; Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Pramipexole; Methylphenidate; Phenelzine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Anhedonia phenotype: PSI (Experimental)
  Interventions: Drug: Pramipexole
- Anhedonia phenotype: CAU (Active Comparator)
  Interventions: Other: Care as usual (CAU) plan
- Cognitive deficits: PSI (Experimental)
  Interventions: Drug: Methylphenidate
- Cognitive deficits: CAU (Active Comparator)
  Interventions: Other: Care as usual (CAU) plan
- Stress sensitivity: PSI (Experimental)
  Interventions: Behavioral: Mindfulness-based Stress Sensitivity Therapy (MBSST)
- Stress sensitivity: CAU (Active Comparator)
  Interventions: Other: Care as usual (CAU) plan
- Anxious distress: PSI (Experimental)
  Interventions: Drug: Phenelzine
- Anxious distress: CAU (Active Comparator)
  Interventions: Other: Care as usual (CAU) plan
- Grief: PSI (Experimental)
  Interventions: Behavioral: Complicated Grief Treatment (CGT)
- Grief: CAU (Active Comparator)
  Interventions: Other: Care as usual (CAU) plan

INTERVENTIONS:
Drug: Pramipexole — CAU plan modified to include a trial of pramipexole.
  Arms: Anhedonia phenotype: PSI
Drug: Methylphenidate — CAU plan modified to include a trial of methylphenidate (or, if contraindicated: guanfacine).
  Arms: Cognitive deficits: PSI
Drug: Phenelzine — CAU plan modified to include a trial of phenelzine (or, if contraindicated: brexpiprazole).
  Arms: Anxious distress: PSI
Behavioral: Mindfulness-based Stress Sensitivity Therapy (MBSST) — CAU plan modified to include a trial of MBSST. MBSST is an individual psychotherapy delivered approximately weekly for 16 sessions.
  Arms: Stress sensitivity: PSI
Behavioral: Complicated Grief Treatment (CGT) — CAU plan modified to include a trial of CGT.
  Arms: Grief: PSI
Other: Care as usual (CAU) plan — Unmodified CAU plan.
  Arms: Anhedonia phenotype: CAU; Anxious distress: CAU; Cognitive deficits: CAU; Grief: CAU; Stress sensitivity: CAU

SUMMARY:
This study aims to assess whether phenotyping-guided intervention selection is superior to intervention selection without phenotyping guidance (i.e., routine clinician and patient judgment regarding treatment selection) for depression.

DETAILED DESCRIPTION:
This study will classify patients seen in the Depression Clinic of the UCSF Department of Psychiatry and Behavioral Sciences into one of five phenotypes (subtypes), including: 1) Anhedonia, 2) Cognitive deficits, 3) Stress sensitivity, 4) Anxious distress, and 5) Grief.

After phenotyping, participants will be randomized to receive phenotype-specific intervention (PSI) or care as usual (CAU).

ELIGIBILITY:
Inclusion Criteria:

* Participant is able to provide informed consent
* English speaker
* 18 years of age or older at time of consent
* Meets DSM-5 criteria for Major Depressive Disorder
* The subject meets eligibility criteria for at least one study phenotype as determined by assessments, imaging and/or clinical judgment.
* PHQ-8 score at baseline of >= 10
* Scheduled for or completed intake in UCSF outpatient psychiatry

Exclusion Criteria:

* Unstable or untreated medical or psychiatric condition based on clinical assessment by investigator(s)
* Significant risk of suicidal or violent behavior as determined by clinical judgement
* In the Investigators' opinion, the subject is not capable of adhering to the protocol requirements, or the subject has a history of poor or suspected poor compliance in clinical research studies, or the subject has a history of poor or suspected poor compliance to antidepressant medication or that study participation is not in their best interest (e.g., different treatment is indicated given their clinical presentation)
* Pregnant or breastfeeding or planning to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptoms - Self-Report 16-Item (QIDS-SR-16) score | Up to 24 weeks after randomization.
  Within-phenotype and across-phenotype contrasts.

SECONDARY OUTCOMES:
Snaith-Hamilton Pleasure Scale (SHAPS) score | Up to 24 weeks after randomization.
  For anhedonia phenotype only.
Clinically Useful Depression Outcome Scale Anxious Distress Specifier Subscale (CUDOS-A) score | Up to 24 weeks after randomization.
  For anxious distress phenotype only.
Generalized Anxiety Disorder 7-item (GAD-7) score | Up to 24 weeks after randomization.
  For anxious distress phenotype only.
Inventory of Complicated Grief (ICG) score | Up to 24 weeks after randomization.
  For grief phenotype only.
Perceived Deficits Questionnaire - Depression (PDQ-D) score | Up to 24 weeks after randomization.
  For cognitive deficits phenotype only.
Patient Health Questionnaire - 8 (PHQ-8) score | Up to 24 weeks after randomization.
  Within-phenotype and across-phenotype contrasts.
WHO Disability Assessment Schedule (WHODAS 2.0) | Up to 24 weeks after randomization.
  Within-phenotype and across-phenotype contrasts.
Quick Inventory of Depressive Symptoms - Self-Report 16-Item (QIDS-SR-16) response | Up to 24 weeks after randomization.
  50% reduction from baseline score. Within-phenotype and across-phenotype contrasts.
Quick Inventory of Depressive Symptoms - Self-Report 16-Item (QIDS-SR-16) remission | Up to 24 weeks after randomization.
  Score < 6. Within-phenotype and across-phenotype contrasts.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D. Krystal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Nancy Friend Pritzker Psychiatry Building, University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No